CLINICAL TRIAL: NCT06531785
Title: Role of Lung Ultrasound in Screening for Interstitial Lung Disease in Patients With Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Assistant Professor of Chest Diseases, Assiut University
Other Study IDs: WGE72024
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Interstitial Lung Disease; Rheumatoid Arthritis
MeSH Terms: conditions — Lung Diseases, Interstitial; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: chest ultrasound — Lung ultrasound to early diagnose ILD among rheumatoid arthritis patients

SUMMARY:
The aim of this observational cross-sectional study is to assess accuracy of Lung Ultrasound to early diagnose ILD among Rheumatoid arthritis patients. Rheumatoid arthritis patients with suggestive history of chest troubles will be evaluated using chest ultrasound and high resolution CT chest to evaluate ability of chest ultrasound to early diagnose ILD among rheumatoid arthritis patients.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) is a common complication of connective tissue disease (CTD) and a leading cause of morbidity and mortality. Thus, early diagnosis and treatment may improve the prognosis of patients with ILD.

High-resolution computed tomography (HRCT) is the gold standard for ILD diagnosis. It can detect the location and type of lesions through its high resolution. Unfortunately, it is hampered by high cost and potential risks associated with radiation exposure, especially for pregnant women.

Accordingly, finding a low-cost, non-invasive, and non-ionizing diagnostic method is necessary for ILD. Lung ultrasound (LUS) has all of these advantages and is an accessible bedside procedure. As a result, it is easily accepted by patients. Over the last 20 years, LUS has mainly been applied in CTD-ILD diagnosis, where it has shown high sensitivity and specificity. The assessment of ILD by LUS is determined by the number of B-lines, which appear as a comet tail signal and originate from the pleural line without fading to the edge of the screen.

The total number of B-lines was found to correlate well with the HRCT score. To assess the number of B-lines, previous studies used various scoring systems by designing different intercostal spaces (LIS), such as 72 LIS, 50 LIS, and 14 LIS. This study aims to assess Lung ultrasound as a screening tool for early interstitial lung disease in connective tissue disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of rheumatoid arthritis and suspicion of interstitial lung disease on history and/ or clinical examination, age > 18 years

Exclusion Criteria:

* Patients who refuse to participate in the study,
* Patients with a history of pulmonary neoplasia or
* Patients with causes of interstitial fluid, such as, heart failure, diastolic dysfunction, asthma or pulmonary edema.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed diagnosis of rheumatoid arthritis and suspicion of interstitial lung disease on history and/ or clinical examination, age > 18 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Number of rheumatoid arthritis patients that can be diagnosed early with Interstitial lung disease. | 1 month
  early diagnosis of Interstitial lung disease among rheumatoid arthritis patients using chest ultrasound versus high resolution computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Waleed MD Gamal Elddin Khaleel, Ass. Prof., Principal Investigator — Assiut University
Locations (1):
- Faculty of Medicine, Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tardella M, Di Carlo M, Carotti M, Filippucci E, Grassi W, Salaffi F. Ultrasound B-lines in the evaluation of interstitial lung disease in patients with systemic sclerosis: Cut-off point definition for the presence of significant pulmonary fibrosis. Medicine (Baltimore). 2018 May;97(18):e0566. doi: 10.1097/MD.0000000000010566. PMID 29718851
- [Background] Ohno Y, Koyama H, Yoshikawa T, Seki S. State-of-the-Art Imaging of the Lung for Connective Tissue Disease (CTD). Curr Rheumatol Rep. 2015 Dec;17(12):69. doi: 10.1007/s11926-015-0546-8. PMID 26483318
- [Background] Tardella M, Gutierrez M, Salaffi F, Carotti M, Ariani A, Bertolazzi C, Filippucci E, Grassi W. Ultrasound in the assessment of pulmonary fibrosis in connective tissue disorders: correlation with high-resolution computed tomography. J Rheumatol. 2012 Aug;39(8):1641-7. doi: 10.3899/jrheum.120104. Epub 2012 Jul 1. PMID 22753655